CLINICAL TRIAL: NCT02346370
Title: PRIMAL STUDY: A Phase 1b, Open-label, Multicenter, Multinational Study of PEGylated Recombinant Human Hyaluronidase (PEGPH20) Combined With Docetaxel (PDoc) in Subjects With Recurrent Previously Treated Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase 1b Study of PEGylated Recombinant Human Hyaluronidase (PEGPH20) Combined With Docetaxel in Subjects With Recurrent Previously Treated Locally Advanced or Metastatic NSCLC
Acronym: PRIMAL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Changing standard of care therapy regimen
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HALO-107-201
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Recurrent, previously treated, locally advanced or metastatic NSCLC (non small cell lung cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — PEGPH20; Docetaxel

STUDY DESIGN:
Intervention Model Description: The study was planned to include a Dose Escalation portion utilizing a standard 3 + 3 dose escalation design. Participants were enrolled sequentially into their assigned dose cohort. The Treatment Period consisted of 21-day treatment cycles with administration of PEGPH20 on Day 1 (doses tested were 1.6, 3.0, and 2.2 ug/kg) and docetaxel (standard dosing 75 mg/m^2 for all participants) on Day 2 of each cycle.
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEGPH20 + Docetaxel (Experimental): PEGylated recombinant human hyaluronidase PH20 (PEGPH20) (1.6, 3.0, or 2.2 micrograms per kilogram (ug/kg)) was administered on Day 1 of each 21-day cycle (every 3 weeks) as an intravenous (IV)-infusion over 10 minutes, approximately 1 milliliter/minute (mL/min) (a window of +2 minutes allowed, i.e., infusion could be 10 to 12 minutes). Docetaxel (75 milligrams/meter squared (mg/m^2)) was administered on Day 2 of each 21-day cycle.
  Interventions: Drug: PEGylated recombinant human hyaluronidase PH20; Drug: Docetaxel

INTERVENTIONS:
Drug: PEGylated recombinant human hyaluronidase PH20
  Other Names: PEGPH20
Drug: Docetaxel
  Other Names: Taxotere

SUMMARY:
A Phase 1b study for participants with Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC) to participate in 1 of 2 portions of this study. The first portion is Dose Escalation in which participants are tested with PEGPH20 at various doses (1.6, 3.0, 2.2 and 2.8 micrograms/kilogram (ug/kg)) in addition to dosing with the standard dose of docetaxel (PDoc) of 75 milligrams/meter squared (mg/m^2) once every 21-day cycle. Based on observations on the safety and tolerability of study treatment from dose escalation cohorts dosed to date (1.6 and 3.0 ug/kg of PEGPH20), two additional dose levels will be tested, 2.2 and 2.8 ug/kg. Up to 30 additional participants may be enrolled to test these dose levels. The second portion of Phase 1b is Cohort Expansion in which the recommended Phase 2 dose (RP2D) of PDoc identified in dose escalation is administered every 21 days to approximately 50 participants with high hyaluronan (HA-high) prospectively measured in their tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Signed, approved Informed Consent.
* Histologically confirmed and documented previously treated Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC), having failed 1 previous platinum chemo regimen for locally advanced or metastatic disease.
* Cohort Expansion: Available archival tumor tissue block or 5-10 unstained, consecutive core biopsy slides from one archival tumor block that meet specific tissue requirements.
* Cohort Expansion: Participants must be determined to be hyaluronidase (HA)-high based on tumor biopsy that meets the requirements noted in the previous inclusion criterion.
* Cohort Expansion: One or more tumors measurable on computed tomography/magnetic resonance imaging (CT/MRI) scan per Response Evaluation Criteria on Solid Tumors (RECIST) v 1.1 (Eisenhauer 2009; Appendix C).
* Participants may have failed a programmed cell death protein 1 (PD-1) or programmed death-ligand 1 (PD-L1) therapy for advanced disease.
* Participants that are known to be epidermal growth factor (EGFR)-activating mutation positive must have received an EGFR inhibitor.
* Participants known to be anaplastic lymphoma kinase (ALK)-fusion/rearrangement mutation positive must have received an ALK inhibitor.
* Most prior therapies and prior targeted therapy are allowed and these specific therapies are detailed in the protocol.
* Life expectancy - =/> 3 months, Eastern Cooperative Oncology Group status = 0 or 1.
* Negative urine or serum pregnancy test within 7 days before Day 1 (first dose of study medication) if female participants is of childbearing potential (WOCBP).
* Men and women agreement to use effective contraceptive method. For WOCBP and for men, agreement to use an effective contraceptive method from the time of screening throughout the study until 1 month for WOCBP or 6 months for men after administration of the last dose of any study medication.
* Specific ranges/levels of Screening labs that are acceptable per protocol.
* Age >/= 18 years.

Exclusion Criteria:

* Previous treatment with docetaxel.
* Failed more than 3 treatment regimens for locally advanced or metastatic NSCLC.
* New York Heart Assoc Class III or IV cardiac disease, myocardial infarction within the past 12 months before screening, or pre-existing atrial fibrillation.
* History of cerebrovascular accident or transient ischemic attack.
* Pre-existing carotid artery disease.
* Previous history of pulmonary embolism or pulmonary embolism found on screening exam.
* No ongoing requirement for corticosteroids
* Active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy at time of screening.
* Known infection with HIV and active infection with hepatitis B or C.
* Known allergy to hyaluronidase or any constituents of docetaxel formulation.
* Current use (within 10 days of day 1) of megestrol acetate.
* Chronic concomitant use of strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, and voriconazole).
* Women currently pregnant or breast feeding.
* Intolerance to dexamethasone, as determined by Investigator.
* History of another primary cancer within the last 3 years that required treatment, with the exception of non-melanoma skin cancer, early stage prostate cancer, or curatively treated cervical carcinoma in situ.
* Any other disease, metabolic dysfunction, physical exam finding, or clinical lab finding that leads to reasonable suspicion of disease that contraindicates the use of an investigational drug that might affect interpretation of results or render subject at high risk for treatment complications.
* In opinion of Investigator, make subject unsuitable for study.
* Hypersensitivity to the active substance or ingredients of PEGPH20 and docetaxel.
* Subject's inability to comply with study and follow-up procedures, as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2016-08-09 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - California Cancer Associates for Research and Excellence (cCare), Encinitas, California
  - California Cancer Associates for Research and Excellence (cCare), Fresno, California
  - Moores UCSD Cancer Center, Clinical Trials Office, San Diego, California
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Rochester, Rochester, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heineman T, Baumgart M, Nanavati C, Gabrail N, Van Wart SA, Mager DE, Maneval DC, Fathallah AM, Sekulovich RE. Safety and pharmacokinetics of docetaxel in combination with pegvorhyaluronidase alfa in patients with non-small cell lung cancer. Clin Transl Sci. 2021 Sep;14(5):1875-1885. doi: 10.1111/cts.13041. Epub 2021 Jul 30. PMID 33982408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 participants were enrolled, of whom 1 participant was not treated due to disease progression prior to treatment and 15 participants received study treatment.
Groups:
- Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel: 1.6 micrograms/kilograms (ug/kg) PEGylated recombinant human hyaluronidase PH20 (PEGPH20) was administered on Day 1 of each 21-day cycle (every 3 weeks) as an intravenous (IV)-infusion over 10 minutes, approximately 1 milliliter/minute (mL/min) (a window of +2 minutes allowed, i.e., infusion could be 10 to 12 minutes). Docetaxel (75 milligrams/meter squared (mg/m^2)) was administered as an IV-infusion on Day 2 of each 21-day cycle.
- Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel: 3.0 ug/kg PEGPH20 was administered on Day 1 of each 21-day cycle (every 3 weeks) as an IV-infusion over 10 minutes, approximately 1 mL/min (a window of +2 minutes allowed, i.e., infusion could be 10 to 12 minutes). Docetaxel (75 mg/m^2) was administered as an IV-infusion on Day 2 of each 21-day cycle.
- Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel: 2.2 ug/kg PEGPH20 was administered on Day 1 of each 21-day cycle (every 3 weeks) as an IV-infusion over 10 minutes, approximately 1 mL/min (a window of +2 minutes allowed, i.e., infusion could be 10 to 12 minutes). Docetaxel (75 mg/m^2) was administered as an IV-infusion on Day 2 of each 21-day cycle.
Period: Overall Study
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Started | 8 | 4 | 4
Completed | 0 | 0 | 0
Not Completed | 8 | 4 | 4
Not completed — Not treated | 1 | 0 | 0
Not completed — Withdrawal of consent | 1 | 0 | 0
Not completed — Death | 1 | 3 | 1
Not completed — Sponsor discontinued study | 5 | 0 | 2
Not completed — Radiologic progression | 0 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel | Total
Number analyzed (Participants) | 7 | 4 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.90) | 57.8 (10.53) | 65.5 (8.10) | 62.6 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 2 | 10
  Male | 1 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 3 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 1 | 0 | 2
  White | 6 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as adverse events (AEs) that occurred during Cycle 1 in the Dose Escalation portion of the study, and deemed by the Investigator as related to study treatment.
Time Frame: Cycle 1 (Day 1 through Day 21) (1 Cycle = 21 days)
Population: The DLT-Evaluable population included all participants who received a full dose of study treatment and completed the initial 21 days of the study after the first dose or who experienced a DLT within the initial 21 days after the first dose and discontinued from the study (if they received a full dose of study drug).
Measure: Number; unit: DLTs
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 7 | 4 | 4
DLTs
  Neutropenia | 0 | 1 | 0
  Gastroenteritis Escherichia coli | 0 | 1 | 0
  Sepsis | 0 | 1 | 0
  Deep vein thrombosis | 0 | 1 | 1

2. Primary Outcome: Number of Participants With the Indicated Type of Adverse Events for PEGPH20 and Docetaxel
Description: Throughout the Treatment Period, the assessment of safety was based on AEs, including deaths, non-serious AEs, and serious adverse events, AEs leading to discontinuation of study treatment, and results of vital sign measurements and clinical laboratory assessments (including hematology, clinical chemistry, coagulation parameters, and urinalysis). Additionally, thromboembolic (TE) events were deemed by the Sponsor as AEs of special interest. AEs and laboratory values were graded for severity using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: From date of first dose until 30 days after the last dose of study treatment, up to approximately 1 year 10 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel: 1.6 ug/kg PEGPH20 was administered on Day 1 of each 21-day cycle (every 3 weeks) as an IV-infusion over 10 minutes, approximately 1 mL/min (a window of +2 minutes allowed, i.e., infusion could be 10 to 12 minutes). Docetaxel (75 mg/m^2) was administered as an IV-infusion on Day 2 of each 21-day cycle.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 7 | 4 | 4
Participants
  AEs greater than or equal to grade 3 | 5 | 4 | 3
  PEGPH20-related AEs | 6 | 4 | 4
  Docetaxel-related AEs | 7 | 4 | 4
  AEs with outcome of death | 0 | 0 | 0
  SAEs | 3 | 3 | 1
  Treatment-related SAEs | 1 | 2 | 1
  AEs leading to discontinuation of study drug | 1 | 1 | 2

3. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of PEGPH20
Time Frame: Cycle 1 of Dose Escalation portion (Cycle 1 = 21 days)
Population: The MTD and RP2D were not established due to early study discontinuation.
Groups:
- PEGPH20 + Docetaxel: PEGPH20 (1.6, 3.0, or 2.2 ug/kg) was administered on Day 1 of each 21-day cycle (every 3 weeks) as an IV-infusion over 10 minutes, approximately 1 mL/min (a window of +2 minutes allowed, i.e., infusion could be 10 to 12 minutes). Docetaxel (75 mg/m^2) was administered as an IV-infusion on Day 2 of each 21-day cycle.
Arm/Group | PEGPH20 + Docetaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1b: Maximum Plasma Concentration (Cmax) of PEGPH20 and Docetaxel
Description: Blood samples were collected from all participants per protocol and analyzed for plasma PEGPH20 concentration using a validated electrochemiluminescence (ECL) immunoassay. Plasma docetaxel concentrations were analyzed using a validated liquid chromatography with tandem mass spectrometry assay (LS-MS/MS). The following blood draw schedule was used, PEGPH20: Cycle 1 Day 1 (C1D1) (predose, 15 minutes (min), 1, 2 to 4, and 24 hours (hr) postdose), C2 and all subsequent Cycles (predose, 1 hr postdose). Docetaxel: C1D2 (30 min after the start of the 1-hr infusion, 30 min post completion of the infusion, 4 to 6 and 24 hr post infusion), C1D3 (24 hr post infusion), C2D2 and C3D2 (30 min after the start of the 1-hour infusion, 30 min post completion of the infusion).
Time Frame: PEGPH20: multiple time points C1D1 and all subsequent Cycles; Docetaxel: multiple time points C1D2, C2D2 and C3D2
Population: Due to early discontinuation of the study, Cmax was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Phase 1b: Minimum Plasma Concentration (Cmin) of PEGPH20 and Docetaxel
Description: Blood samples were collected from all participants per protocol and analyzed for plasma PEGPH20 concentration using a validated ECL immunoassay. Plasma docetaxel concentrations were analyzed using a validated liquid chromatography with LS-MS/MS. The following blood draw schedule was used, PEGPH20: C1D1 (predose, 15 min, 1, 2 to 4, and 24 hr postdose), C2 and all subsequent Cycles (predose, 1 hr postdose). Docetaxel: C1D2 (30 min after the start of the 1-hr infusion, 30 min post completion of the infusion, 4 to 6 and 24 hr post infusion), C1D3 (24 hr post infusion), C2D2 and C3D2 (30 min after the start of the 1-hour infusion, 30 min post completion of the infusion).
Time Frame: PEGPH20: multiple time points C1D1 and all subsequent Cycles; Docetaxel: multiple time points C1D2, C2D2 and C3D2
Population: Due to early discontinuation of the study, Cmin was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Phase 1b: Time to Maximum Plasma Concentration (Tmax) of PEGPH20 and Docetaxel
Description: as for outcome 5
Time Frame: PEGPH20: multiple time points C1D1 and all subsequent Cycles; Docetaxel: multiple time points C1D2, C2D2 and C3D2
Population: Due to early discontinuation of the study, Tmax was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Phase 1b: Terminal Half-life (t1/2) of PEGPH20 and Docetaxel
Description: as for outcome 5
Time Frame: PEGPH20: multiple time points C1D1 and all subsequent Cycles; Docetaxel: multiple time points C1D2, C2D2 and C3D2
Population: Due to early discontinuation of the study, t1/2 was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve for PEGPH20 and Docetaxel
Description: as for outcome 5
Time Frame: PEGPH20: multiple time points C1D1 and all subsequent Cycles; Docetaxel: multiple time points C1D2, C2D2 and C3D2
Population: Due to early discontinuation of the study, the AUC was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Phase 1b: Volume of Distribution (Vd) of PEGPH20 and Docetaxel
Description: as for outcome 5
Time Frame: PEGPH20: multiple time points C1D1 and all subsequent Cycles; Docetaxel: multiple time points C1D2, C2D2 and C3D2
Population: Due to early discontinuation of the study, Vd was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Phase 1b: Clearance (CL) of PEGPH20 and Docetaxel
Description: as for outcome 5
Time Frame: PEGPH20: multiple time points C1D1 and all subsequent Cycles; Docetaxel: multiple time points C1D2, C2D2 and C3D2
Population: Due to early discontinuation of the study, CL was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR = complete response + partial response (CR + PR)
Time Frame: From date of treatment start until disease progression or up to data cutoff date (30 Nov 2016), for up to approximately 1 year 9 months
Population: Due to early discontinuation of the study, ORR was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Disease Control Rate (DCR)
Time Frame: as for outcome 11
Population: Due to early discontinuation of the study, DCR was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Duration of Response (DoR)
Time Frame: From date of first CR or PR until the date of first documentation of disease progression or date of death, assessed up to data cutoff date (30 Nov 2016)
Population: Due to early discontinuation of the study, DoR was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: From date of treatment start until date of first documentation of progressive disease or death from any cause, assessed up to 1 year 9 months
Population: Due to early discontinuation of the study, PFS was not assessed.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose until 30 days after the last dose of study drug, up to approximately 1 year 10 months.
Description: Treatment-emergent adverse events (TEAEs) and serious adverse events were reported. Adverse event severity was assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03. The Safety Population was evaluated and included all participants who received at least one dose of study treatment.
Arm/Group | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel
All-Cause Mortality (participants affected / at risk) | 1/7 | 3/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 3/7 | 3/4 | 1/4
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel (N=7) | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel (N=4) | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel (N=4)
Pneumonia (Infections and infestations) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 1.6 ug/kg PEGPH20 + Docetaxel (N=7) | Cohort 2: 3.0 ug/kg PEGPH20 + Docetaxel (N=4) | Cohort 3: 2.2 ug/kg PEGPH20 + Docetaxel (N=4)
Fatigue (General disorders) | 6 | 3 | 4
Oedema peripheral (General disorders) | 3 | 0 | 1
Pyrexia (General disorders) | 4 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Candida infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 2
Cushingoid (Endocrine disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was discontinued early by the Sponsor during the Dose Escalation Period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other